CLINICAL TRIAL: NCT03113214
Title: Phase I Study of PET/CT-directed Hyperfractionated Radiation Dose Escalation With Concurrent Weekly Carboplatin and Paclitaxel in Esophageal Cancer
Brief Title: PET/CT-directed Hyperfractionated Radiation Dose Escalation in Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chen tingfeng, director, department of radiation, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGH201713
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2018-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- radiochemotherapy 1 (Experimental): Patients will be treated with radiation therapy 57.2 Gy.
  Interventions: Radiation: radiochemotherapy 1
- radiochemotherapy 2 (Experimental): Patients will be treated with radiation therapy 64.4 Gy.
  Interventions: Radiation: radiochemotherapy 2
- radiochemotherapy 3 (Experimental): Patients will be treated with radiation therapy 71.6 Gy.
  Interventions: Radiation: radiochemotherapy 3
- radiochemotherapy 4 (Experimental): Patients will be treated with radiation therapy 78.8 Gy.
  Interventions: Radiation: radiochemotherapy 4
- radiochemotherapy 5 (Experimental): Patients will be treated with radiation therapy 86 Gy.
  Interventions: Radiation: radiochemotherapy 5
- radiochemotherapy 6 (Experimental): Patients will be treated with radiation therapy 93.2 Gy.
  Interventions: Radiation: radiochemotherapy 6

INTERVENTIONS:
Radiation: radiochemotherapy 1 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 7.2 Gy at 1.2 Gy/Fx/bid to residual tumor volume as defined by PET/CT; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2, weekly; paclitaxel, 45-50 mg/m2, weekly
  Other Names: concurrent radiochemotherapy 1
  Arms: radiochemotherapy 1
Radiation: radiochemotherapy 2 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 14.4 Gy at 1.2 Gy/Fx/bid to residual tumor volume as defined by PET/CT;
  Other Names: concurrent radiochemotherapy 2
  Arms: radiochemotherapy 2
Radiation: radiochemotherapy 3 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 21.6 Gy at 1.2 Gy/Fx/bid to residual tumor volume as defined by PET/CT;
  Other Names: concurrent chemoradiotherapy regimen 3
  Arms: radiochemotherapy 3
Radiation: radiochemotherapy 4 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 28.8 Gy at 1.2 Gy/Fx/bid to residual tumor volume as defined by PET/CT;
  Other Names: concurrent chemoradiotherapy regimen 4
  Arms: radiochemotherapy 4
Radiation: radiochemotherapy 5 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 36 Gy at 1.2 Gy/Fx/bid to residual tumor volume as defined by PET/CT;
  Other Names: concurrent chemoradiotherapy regimen 5
  Arms: radiochemotherapy 5
Radiation: radiochemotherapy 6 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 43.2 Gy at 1.2 Gy/Fx/bid to residual tumor volume as defined by PET/CT;
  Other Names: concurrent chemoradiotherapy regimen 6
  Arms: radiochemotherapy 6

SUMMARY:
The goal of this study is to find the maximum tolerable dose of radiation that can be delivered with concurrent chemotherapy (carboplatin & paclitaxel) in patients with esophageal cancer.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy is the standard of care for esophageal cancer based on the results of phase III randomised trials. The current standard radiation therapy dose has remained 50 Gy at -2 Gy/fraction for decades.However, locoregional control remain problematic, with 25% of patients having persistence and 20% relapse of locoregional disease following the combined modality approach. New regimen is urgently needed for improving localregional control and survival.Investigators hypothesize that hyperfractionated radiation dose escalation to residual tumor volumes after standard chemoradiotherapy as defined by positron emission tomography (PET) /computed tomography (CT) would improve local control and overall survival while reducing the acute and late normal tissue toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed primary squamous cell carcinoma of the esophagus
2. Age 1 8-75.
3. Patients must be deemed unresectable disease or patient is not deemed operable due to medical reasons.
4. Patients with distant metastasis and life expectancy >/= 3 months are eligible.
5. Zubrod performance status 0 to 2
6. No prior radiation to the thorax that would overlap with the current treatment field.
7. Patients with nodal involvement are eligible
8. Adequate bone marrow, renal and hepatic functions as assessed by the following: Hemoglobin >/= 10.0 g/dl, Platelet count >/= 1 00,000/mm^3,absolute granulocyte count (AGC) ≥2 × 10^9 cells/L,bilirubin and Aspartate transaminase ≤1.5 ×upper limit of normal (ULN), Creatinine </=1 .5 times ULN.
9. A signed informed consent must be obtained prior to therapy. 1 0. Induction chemotherapy is allowed

Exclusion Criteria:

1. The presence of a fistula.
2. Prior radiotherapy that would overlap the radiation fields.
3. gastroesophageal junction cancer.
4. Uncontrolled concurrent illness including, but not limited to: Chronic 5.Obstructive Pulmonary Disease(COPD) exacerbation or other respiratory illness, serious uncontrolled infection, symptomatic congestive heart failure (CHF),unstable angina pectoris, uncontrolled hypertension,or psychiatric illness/social situations that would limit compliance with the study requirements.

6.Known hypersensitivity to paclitaxel. 7.Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.

Acquired Immune Deficiency Syndrome. 8.Conditions precluding medical follow-up and protocol compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 1 year
  Maximum Tolerated Dose is defined as CTCAE 4 grade 3 acute radiation-related toxicity

SECONDARY OUTCOMES:
Time to Local Failure | 2 years
  Local control will be assessed radiographically using endoscopy with biopsy and a positron emission computed tomography-CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Tingfeng Chen, MD, Study Director — the ethic committee of shanghai genernal hospital
Locations (1):
- Shanghai Genernal Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No